CLINICAL TRIAL: NCT06178809
Title: Clinical Research on Dynamic Monitoring MRD Via Plasma ctDNA Predicting Postoperative Recurrence and Progression After Systemic Therapy of Hepatocellular Carcinoma
Brief Title: Clinical Research on Dynamic Monitoring MRD Via Plasma ctDNA After Systemic Therapy of Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Singlera Genomics Inc. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYS-2021002
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; MRD; ctDNA; Mutation; Methylation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to combine biomarker characteristic atlas and ctDNA detection technology to establish a precise standard scheme for minimal residual diagnosis of liver cancer after surgery and systemic treatment.

DETAILED DESCRIPTION:
This study is a prospective, single-blind, randomized, controlled, single-center study. The patients with liver cancer are recruited after surgery or systemic treatment. Intraoperative cancer and para-cancer tissues of surgical patients are collected, and peripheral blood of all patients after multiple follow-up visits before and after treatment are also collected. The established detection method and model are used to detect blood ctDNA of patients with liver cancer after treatment, and the follow-up data are collected to observe the correlation between the genomic characteristics of plasma at multiple follow-up points after treatment and the recurrence or progression after treatment. The sensitivity and specificity of ctDNA detection method is calculated to predict the risk of relapse or progression after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old (including 80 years old), gender is not limited;
2. Patients diagnosed with primary HCC;
3. ECOG score ≤1;
4. no previous malignant tumors, including liver cancer;
5. Before blood collection, the patient had not received any treatment related to liver cancer, including surgery, transplantation, radiotherapy, chemotherapy, etc.;
6. Survival period of ≥3 years as initially assessed by researchers;
7. Those who are fully aware of this study and voluntarily sign the informed consent.

Exclusion Criteria:

1. Patients diagnosed with esophageal cancer, gastric cancer, colorectal cancer, lung cancer, pancreatic cancer, breast cancer and other malignant tumors;
2. Patients who have received major surgical treatment such as blood transfusion or transplantation within 3 months;
3. Participate in other interventional clinical investigators within 3 months;
4. Pregnant or lactating women;
5. Patients with autoimmune diseases, genetic diseases, mental disorders/disabilities, substance abuse and other diseases deemed unsuitable for participation in the study by the researchers;
6. Poor compliance, according to the judgment of the researcher can not complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-80 years old primary hepatocellular carcinoma patients in Zhongshan hospital, Shanghai, China
Sampling Method: Probability Sample
Enrollment: 475 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of plasma ctDNA mutation and methylation model to predict disease-free survival (DFS) or progression-free survival (PFS) in patients with primary hepatocellular carcinoma after treatment | 2 years
  Plasma ctDNA mutation and methylation are detected after treatment in patients with primary hepatocellular carcinoma who underwent hepatectomy or systemic therapy. Clinical information of disease-free survival (DFS) or progression-free survival (PFS) is collected to explore the predictive effect of plasma ctDNA mutation and methylation status on the prognosis of primary hepatocellular carcinoma after treatment.
The advance time of ctDNA dynamic detection compared with AFP+ imaging in monitoring of primary hepatocellular carcinoma recurrence or progression | 6 months
  Patients with primary hepatocellular carcinoma who underwent hepatectomy or systemic therapy are followed up regularly after treatment. During follow-up, plasma ctDNA test results, traditional tumor marker AFP and imaging evaluation data are collected. Mutations and methylation of plasma ctDNA are detected. All the data is analyzed to explore the advance time of dynamic detection of plasma ctDNA mutation and methylation in monitoring recurrence or progression of primary hepatocellular carcinoma compared with AFP+ imaging monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Fudan university Zhongshan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided